CLINICAL TRIAL: NCT05704270
Title: The Efficacy of Computerized Cognitive Training in Patients With Hypertension and Cognitive Impairment, no Dementia: a Randomized Controlled Trial
Brief Title: Computerized Cognitive Training to Protect Cognitive Function Among Hypertension Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Wispirit Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Chang sheng Ma, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022BFAZ01
Record Dates: First submitted 2023-01-09; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Mild Cognitive Impairment; Hypertension
Keywords: Cognitive training; Digital health; Hypertension
MeSH Terms: conditions — Cognitive Dysfunction; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive cognitive training (Experimental): This arm is the intervention arm. Participants randomized to this arm will use a tablet to receive the multi-domain adaptive cognitive training, which will be delivered 30 minutes at least 5 times a week for 12 weeks.
  Interventions: Behavioral: Multi-domain adaptive cognitive training
- Active control (Active Comparator): This arm is the control arm. Participants randomized to this arm will use the same tablet to receive the cognitive training of low difficulty level with no adaptive change. The intervention dosage will be the same, which is 30 minutes each time, at least 5 times a week for 12 weeks.
  Interventions: Behavioral: Basic cognitive training with no difficulty change

INTERVENTIONS:
Behavioral: Multi-domain adaptive cognitive training — The multi-domain adaptive cognitive training covers seven aspects of fundamental cognitive function, including sensory perception, cognitive flexibility, attention, memory, language, logic calculation, and emotion recognition and management. A self-adaptive algorithm is embedded in the tablet-based cognitive training platform, which will help deliver suitable tasks at the right difficulty level for each participant according to their personal profile and real-time performance. The intervention dosage is 30 minutes per time, 5 times a week.
  Arms: Adaptive cognitive training
Behavioral: Basic cognitive training with no difficulty change — The basic cognitive training for the control arm will also be delivered via a tablet. The training tasks will be fixed at a primary difficulty level without adaptive algorithm. The intervention dosage is also 30 minutes per time, 5 times a week.
  Arms: Active control

SUMMARY:
Hypertension is an risk factor for cognitive impairment. The primary objective of this study is to evaluate the efficacy of 12-week computerized cognitive training in people with hypertension and mild cognitive impairment. The researchers will further investigate the long-term effects of cognitive training by prolonging the intervention for 24 weeks among a randomly selected sub-group.

DETAILED DESCRIPTION:
This study is a double-blinded, randomized controlled trial. A total of 200 hypertension patients with mild cognitive impairment will be recruited to participate in this study after screening. These patients will be randomized to two arms under masking. The intervention arm will receive multi-domain adaptive cognitive training using a tablet. The control arm will receive an active control treatment and use the same tablet to receive the cognitive training tasks with weak difficulty change. Both arms will receive the same intervention dosage for 12 weeks, 5 times a week, and 30 minutes per time. After the 12-week intervention, the intervention arm will be re-randomized into two groups. One group will stop their intervention at 12 weeks; the other group will continue to receive the multi-domain adaptive cognitive training till the 24-week follow-up assessment.

The neuro-psychological assessment will be administered at baseline, 12-week, and 24-week assessments for all participants. The structural and functional MRI will be administered at baseline, 12 weeks, and 24 weeks to evaluate the effect of cognitive training on brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 60 years;
2. Completed 6 or more years of education;
3. Untreated or under treatment hypertension;
4. Complaint of memory decline within 1 year;
5. Global cognitive score measured by the Montreal Cognitive Assessment is below 26;
6. Agree to receive cognitive function evaluation, randomization, and follow-up investigation as required;

Exclusion Criteria:

1. Unable to complete cognitive function evaluation due to vision, hearing, and other problems;
2. Have been diagnosed of dementia or MMSE score ≤ 20;
3. Unable to use the cognitive training equipment after 2 times instructions;
4. Alcohol abuse or taking drugs that could affect cognitive function (antihistamines, antipsychotics);
5. Diabetes patients;
6. Moderate to severe decrease in glomerular filtration rate (eGFR<30 ml/min /1.73m2);
7. Systolic blood pressure ≥180 mmHg or/and diastolic blood pressure ≥110 mmHg; or orthostatic hypotension (defined as the third standing SBP<100mmHg);
8. History of cardiovascular events or hospitalization due to cardiovascular diseases in the last 3 months;
9. Planned to receive coronary intervention, atrial fibrillation ablation or cardiac surgery within 6 months; or have received these intervention strategies in the last 3 months;
10. Symptomatic heart failure or left ventricular ejection fraction <50%；
11. Atrial fibrillation confirmed by ECG with marked and severe onset of symptoms;
12. A history of stroke, or head injury in the last 6 months; past history of brain tumor or neurosurgery;
13. Past history of Parkinson's disease, Alzheimer's disease, schizophrenia, and epilepsy;
14. Have Ever undergone surgery under general anesthesia in the last three months;
15. Severe hepatic impairment or in critical condition patients with very poor prognosis whose expected survival is less than 6 months; or diagnosed of malignant tumor other than non-melanoma skin cancer in the last 2 years;
16. Contradictions for MRI examination: such as metal implantation, claustrophobia, etc.;
17. Unable to obtain an informed consent or currently taking part in other clinical trials

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Global cognitive function change measured by BCAT in 12 weeks | 12 weeks after randomization
  The proportion of patients whose global cognitive function improves 0.67SD compared to the baseline cognitive function measured by Basic Cognitive Ability Test (BCAT). BCAT is a set of neuropsychological battery tests which was designed to measure global cognitive fucntion and cognitive function of sub-domains. Higher scores of BCAT means a better global cognitive function.

SECONDARY OUTCOMES:
Global cognitive function change measured by BCAT in 24 weeks | 24 weeks after randomization
  The proportion of patients whose global cognitive function improves 0.67SD compared to the baseline cognitive function at 24 weeks measured by Basic Cognitive Ability Test(BCAT).
Sub-domain cognitive function improvement including memory, attention, and execution memory | 12 weeks, 24 weeks after randomization
  The proportion of patients whose sub-domain cognitive function, including attention, memory, execution function improves measured by the individual capability test in BCAT.
Cognitive score change | 12 weeks, 24 weeks after randomization
  Mean change from baseline in global cognitive function score measured by basic cognitive ability test (BCAT) at 12 weeks and 24 weeks.
Self-efficacy score | 12 weeks, 24 weeks after randomization
  Mean change from baseline in self-efficacy score measured by the General Self-Efficacy Scale at 12 weeks, and 24 weeks
Quality of life score | 12 weeks, 24 weeks after randomization
  Mean change from baseline in the patient's quality of life score measured by EQ-5D-3L at 12 weeks and 24 weeks.
Anxiety score | 12 weeks, 24 weeks after randomization
  Mean change from baseline in the patient's anxiety score at 12 weeks and 24 weeks. Anxiety status will be measured by GAD-7 questionnaire. Higher score of GAD-7 scale represents more anxiety status.
Depression score | 12 weeks, 24 weeks after randomization
  Mean change from baseline in the patient's depression score at 12 weeks and 24 weeks. Depression status will be measured by PHQ-9 questionnaire. Higher score of PHQ-9 scale represents more depression status.

CONTACTS AND LOCATIONS:
Overall Officials: Chang sheng Ma, Principal Investigator — Beijing Anzhen Hospital
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Beijing
  - Ruijing Hospital, Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kong Y, Guo QH, Zhou L, He L, Zeng Y, Du X, Dong JZ, Jiang C, Wang JG, Ma CS. Digital computerised cognitive training for preventing cognitive decline among hypertensive patients: a study protocol for a multicentre randomised controlled trial (DELIGHT trial). BMJ Open. 2024 Feb 29;14(2):e079305. doi: 10.1136/bmjopen-2023-079305. PMID 38423771